CLINICAL TRIAL: NCT06633757
Title: A Phase 1b, Open-label, Study of RCT1100 in Adults With Primary Ciliary Dyskinesia Caused by Pathogenic Mutations in the DNAI1 Gene to Measure Mucociliary Clearance and Other Measures of Pharmacodynamic Activity
Brief Title: Study of Inhaled RCT1100 in Adults With PCD Caused by Pathogenic Mutations in the DNAI1 Gene to Measure Mucociliary Clearance
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ReCode Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCT1100-103
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Primary Ciliary Dyskinesia (PCD)
Keywords: Primary ciliary Dyskinesia; PCD; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PCD Participants (Experimental): RCT1100 mRNA therapy supplied to eligible participants with Primary Ciliary Dyskinesia caused by disease-causing mutations in the DNAI1 gene
  Interventions: Drug: RCT1100

INTERVENTIONS:
Drug: RCT1100 — mRNA therapy supplied as varying dose strengths administered via oral inhalation using nebulizer

SUMMARY:
This is a multi-dose study with RCT1100 and is designed to provide safety, tolerability and preliminary efficacy data for future clinical studies.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the impact of multiple doses of inhaled RCT1100, administered via nebulizer, on MCC with adult participants with Primary Ciliary Dyskinesia caused by pathogenic mutations in the DNAI1 Gene.

ELIGIBILITY:
Major Inclusion Criteria:

* The participant is a male or female, 18 to 75 years of age, inclusive, at the time of consent.
* Participant has disease-causing (pathogenic and/or likely pathogenic) mutations in the DNAI1 gene.
* The participant has a percent predicted forced expiratory volume in 1 second (FEV1pp) of at least 40% predicted.

Exclusion Criteria:

* History or presence of clinically significant medical, surgical, clinical laboratory, or psychiatric condition or disease.
* History of cancer, with exception of adequately treated basal cell or squamous cell carcinoma of the skin.
* Predisposition to bleeding or clinically meaningful hemorrhagic event in the 12 months prior
* Medically significant hemoptysis.
* Anticoagulation therapy for the treatment of a pulmonary embolus or has had a pulmonary embolus in the last 6 months of screening.
* Active tuberculosis infection.
* 12-lead ECG with QT interval >450 msec (or >480 msec for BBB)
* Laboratory abnormalities in clinical laboratory tests at screening:

  1. Serum creatinine level
  2. Total bilirubin, aspartate aminotransferase or alanine aminotransferase values
  3. Hematological or coagulation values outside the normal reference range
* Any medical history of disease that has the potential to cause a rise in total bilirubin over the ULN.
* COVID-19 infection within 4 weeks of Screening or receipt of COVID-19 vaccine within 2 weeks prior to first dose of RCT1100.
* Receipt of vaccine with live virus, attenuated live virus, or live viral components within 2 weeks prior to first dose of RCT1100 or to receive these vaccines during treatment or within 8 weeks of completion of study treatment.

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To Determine the impact of multiple doses of RCT1100 on MCC | Baseline through Week 12
  The Change in Mucociliary and Cough Clearance through 1 hour after radiotracer administration by either the albumin-based PRMC or sulfur-colloid technique

CONTACTS AND LOCATIONS:
Overall Officials: John Matthews, MBBS, MCRP, PhD, Study Chair — ReCode Therapeutics, Inc.; Heymut Omran, MD, Principal Investigator — University Hospital Muenster; Kim G Nielsen, Dr Med Sci, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- UNC, Chapel Hill, North Carolina, United States
- Copenhagen University Hospital - Rigshospitalet, Copenhagen, Denmark
- Münster University Hospital, Albert-Schweitzer-Campus 1, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No